CLINICAL TRIAL: NCT04380311
Title: Precision Pharmacokinetic-Guided Tacrolimus Dosing to Improve Pediatric Heart Transplant Outcomes
Brief Title: Precision Guided Tacrolimus Dosing in Pediatric Heart Transplant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joseph Rower, Research Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00124800; K01HL148402 (NIH)
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Heart Transplant Failure and Rejection
Keywords: Tacrolimus, Pediatrics
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Precision Tacrolimus (Experimental): Participants in this arm of the study will have their tacrolimus dose determined using a precision medicine decision support software tool. The participant's transplant physician will consider the recommended dose from the decision support tool in combination with the physician's expertise and experience to determine the proper tacrolimus dose for the participant.
  Interventions: Device: Tacrolimus Dosing Support Tool

INTERVENTIONS:
Device: Tacrolimus Dosing Support Tool — The tacrolimus dosing support tool is based on a population pharmacokinetic model that incorporates patient specific factors including age, renal function, and concomitant medications.
  Other Names: Tacrolimus

SUMMARY:
Immunosuppressive therapy is required to prevent organ rejection, however, dosing of immunosuppressive agents is complicated by patient-specific differences impacting the body's absorption and elimination of these agents. The goal of this research proposal is to clinically validate an innovative precision medicine strategy for dosing the immunosuppressant tacrolimus in pediatric heart transplant, which will in turn lead to improvements in long-term transplant survival outcomes. The strategy and techniques used in this project can be extended to improve drug therapy across multiple pediatric diseases requiring chronic therapy.

DETAILED DESCRIPTION:
Of the more than 400 children annually receiving a heart transplant, the likelihood that the child dies within five years (25%) is equivalent to the potential that the child lives >20 years post-transplant. The success of the transplant, and thus long-term survival of the child, is well known to correlate with achieving adequate immunosuppression to prevent rejection, especially in the period immediately following transplant. Attaining adequate immunosuppression is complicated by several factors, many of which impact the pharmacokinetics (PK) of the immunosuppressive agent. These factors include age of the patient, renal and hepatic function, concomitant medications, patient genetics, and the time post-transplant. Frequent, invasive drug monitoring is used clinically to assess how these factors impact an individual child's PK, and in turn the dose required to achieve and maintain adequate immunosuppression. However, this empirical "guess and check" approach often results in the child spending substantial time receiving immunosuppressive therapy that is either ineffective or unsafe, decreasing the longevity of the transplant organ and thus, long-term patient survival. A more desirable approach would be to guide dosing using a precision medicine approach, wherein patient specific factors are used a priori to predict the dose most likely to achieve adequate immunosuppression. Developing a precision medicine platform for immunosuppression following pediatric heart transplant has the potential to not only improve outcomes in heart transplant recipients, but across all transplant types. This proposal aims to: 1) determine the impact of CYP3A5 genetic variation on tacrolimus concentrations in children, 2) prospectively validate the clinical utility of a PK-guided precision medicine platform in pediatric heart transplant patients receiving tacrolimus-based immunosuppression; and 3) identify and correlate biomarkers of transplant outcomes and tacrolimus safety/effect with the PK of tacrolimus, in order to establish the tacrolimus concentrations required for safe and effective immunosuppression in pediatric heart transplant recipients. The overall objective of this study is to improve the long-term survival of children with heart transplant via optimization of the child's immunosuppressive therapy. Importantly, the interdisciplinary nature of this mentored research proposal will facilitate my progress towards an independent career developing precision medicine tools to improve health outcomes in children.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 6 months and less than 18 years.
2. Received heart transplant for congenital heart malformation or cardiomyopathy.

Exclusion Criteria:

1. Unwillingness to complete study procedures.
2. Significant comorbidity that would prevent study completion.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to target concentration attainment | Within 6 weeks following transplant
  Target attainment will be defined concentrations within the target range (10-15 ug/L) and no dose modifications for 3 consecutive days. Time to target concentration in the intervention arm will be compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Rower, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rower JE, Stockmann C, Linakis MW, Kumar SS, Liu X, Korgenski EK, Sherwin CMT, Molina KM. Predicting tacrolimus concentrations in children receiving a heart transplant using a population pharmacokinetic model. BMJ Paediatr Open. 2017;1(1):e000147. doi: 10.1136/bmjpo-2017-000147. Epub 2017 Nov 22. PMID 29177199